CLINICAL TRIAL: NCT04100499
Title: Evaluation of Adjunctive Use of EndoAnchors During of After EVAR and TEVAR
Brief Title: Evaluation of Adjunctive EndoAnchors for EVAR and TEVAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Andrés Reyes Valdivia, Principal Investigator, Hospital Universitario Ramon y Cajal
Other Study IDs: 187/19
Record Dates: First submitted 2019-09-19; First posted 2019-09-24 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Aortic Aneurysm; Thoracic Aortic Aneurysm
Keywords: Endoanchors; EVAR; TEVAR
MeSH Terms: conditions — Aortic Aneurysm; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: ESAR (Endosutured Aneurysm Repair) — EndoAnchors adjunctive therapy for EVAR and TEVAR

SUMMARY:
EndoAnchors (Heli-FX device, Medtronic, Santa Rosa) have beed described to improve fixation (mimicking an open surgical anastomosis) during or after EVAR/TEVAR.

The investigators want to describe the outcomes of all consecutive patients treated with this device (retrospective and prospective data - observational study)

DETAILED DESCRIPTION:
EndoAnchors (Heli-FX device, Medtronic, Santa Rosa) have beed designed to improve the Endovascular aortic repair. This device is described to mimic an open surgical anastomosis during or after EVAR/TEVAR.

The investigators want to describe the outcomes of all consecutive patients treated with this device (retrospective and prospective data - observational study), these outcomes will be described in terms of type IA Endoleaks, migration and sac regression.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with adjunctive use of EndoAnchors during or after EVAR and TEVAR

Exclusion Criteria:

* Patients that don't want te receive any repair for their disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with abdominal or thoracic aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-11-19 (Estimated)

PRIMARY OUTCOMES:
Rate of participants with type IA Endoleaks | Three years
  Absence of type IA Endoleaks during follow-up

SECONDARY OUTCOMES:
Rate of participants with Endograft Migration | Three years
  Analysis of Endograft migration during follow-up
Rate of participants with Sac regression | Three years
  Analysis of Sac regression during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andres Reyes Valdivia, Consultant, Principal Investigator — Vascular Surgery Department
Locations (1):
- Vascular Surgery Department, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reyes Valdivia A, Duque Santos A, Pitoulias G, Aracil Sanus E, Ocana Guaita J, Gandarias Zuniga C. Predictors of inadequate EndoAnchors aortic wall penetration for the Endosutured therapy in hostile neck patients. J Cardiovasc Surg (Torino). 2020 Dec;61(6):738-744. doi: 10.23736/S0021-9509.20.11248-5. Epub 2020 Jun 19. PMID 32558525
- [Background] Reyes Valdivia A, Busto Suarez S, Duque Santos A, Zanabili Al-Sibbai AA, Gandarias Zuniga C, Chaudhuri A. Evaluation of EndoAnchor Aortic Wall Penetration After Thoracic Endovascular Aortic Repair. J Endovasc Ther. 2020 Apr;27(2):240-247. doi: 10.1177/1526602820907564. PMID 32186262
- [Derived] Reyes Valdivia A, Milner R, Heijmen R, Riambau V, Rousseau H, Tinelli G, Kotelis D, Zanabili Al-Sibbai AA, Pitoulias G, Zuniga CG, de Beaufort HWL, Panagiotis D, Chaudhuri A. Mid-term outcomes of the use of endoanchors during thoracic endovascular aortic repair in multicentre analysis. Vascular. 2023 Jun;31(3):455-462. doi: 10.1177/17085381221076320. Epub 2022 Feb 27. PMID 35225085
- [Derived] Reyes Valdivia A, Chaudhuri A, Milner R, Pratesi G, Reijnen MM, Tinelli G, Schuurmann R, Barbante M, Babrowski TA, Pitoulias G, Tshomba Y, Gandarias C, Badawy A, de Vries JP. Endovascular aortic repair with EndoAnchors demonstrate good mid-term outcomes in physician-initiated multicenter analysis-The PERU registry. Vascular. 2022 Feb;30(1):27-37. doi: 10.1177/1708538121992596. Epub 2021 Feb 10. PMID 33568007